CLINICAL TRIAL: NCT04775927
Title: Evaluation of the Effectiveness of WEB-Based Marriage Preparation Training Provided to Premarital Couples
Brief Title: Pre-marital Internet-based Sexual and Reproductive Health Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ebru İnan Kırmızıgül (Other)
Responsible Party: Sponsor-Investigator, Ebru İnan Kırmızıgül, Principal Investigater, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Saglik Bilimleri Enstitüsü
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Internet-Based Intervention; Health Knowledge, Attitudes, Practice
Keywords: Sex Education; Online Education
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: There will be ywo group. One is interventional group; other is control group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The volunteer and the researcher (caregiver) before agreeing to participate in the study will not know which group they will be in. After accepting the research, the participant and the researcher will know who will be in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education group (Experimental): marriage preparation training
  Interventions: Other: education
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: education — premarital education
  Arms: education group

SUMMARY:
This research; It is carried out to investigate the effects of Web-based marriage preparation training given to couples applying for marriage on sexual health-reproductive health knowledge, marital adjustment and sexual satisfaction of newly married couples.

DETAILED DESCRIPTION:
Study Group Universe The universe of the study consists of couples living in Ankara who have decided to get married and applied to Çankaya Municipality Marriage Office and / or Altındağ Municipality Marriage Office.

Sample of the Study Group With type I error of 0.05 and 80% power, the minimum number of individuals required to determine the difference in numerical values for the groups at d = 0.50 effect width (medium effect width was taken in the absence of a priori information) was determined as 128 in total. This number will be equally distributed among the groups. Considering the losses that may occur, it is planned to work with at least 50 pairs in the groups. (The sample size and power calculation required for the study was done using the program G * Power, Ver. 3.0.10, Universität Kiel, Germany, http://www.psycho.uni-duesseldorf.de/aap/projects/gpower/)

Consent of couples who apply for marriage will be obtained with an informed voluntary consent form.

Couples who meet the sampling criteria at least 2 months before the wedding / wedding day will be included in the study.

Randomization will be made in determining the training and control groups in the study.

In the first stage, an introductory information form and sexual health-reproductive health knowledge test will be applied face to face to the control group. The introductory information form includes socio-demographic characteristics, characteristics related to marital life, characteristics of sexual and reproductive health and sexual health-reproductive health education.An introductory brochure will be given to the intervention group and the WEB site will be introduced. Introductory information form and sexual health-reproductive health information test will be applied to the intervention group based on WEB.

In the second stage, WEB-based marriage preparation training will be given to the intervention group. The training program is planned in two modules. The first module will include communication and problem solving, while the second module will include sexual health, reproductive health, contraception methods, sexually transmitted infections and domestic violence. Each training topic will be in the form of a 20-minute video narration and will be planned for 2 weeks in total. Participants will be able to benefit from the trainings 24 hours a day, 7 days a week. It will be ensured that the trainings are completed before the wedding. In the second stage, no intervention is applied to the control group. One month after the intervention group got married, the sexual and reproductive health knowledge test will be applied again.

In the third stage, 4 months after marriage, sexual health-reproductive health knowledge test, marital adjustment scale, sexual satisfaction scale and sexual self-efficacy scale will be applied to the intervention group. 4 months after marriage, the data of the marital adjustment scale, sexual satisfaction scale and sexual self-efficacy scale will be obtained from the control group via e-mail or phone.

Evaluation of Data:

The compatibility of the continuous variables to be obtained within the scope of the study to the normal distribution will be examined with the Shapiro-Wilk test. While mean ± standard deviation is used in the representation of descriptive statistics related to the variables that conform to the normal distribution, the median (Interquartile Width - MPI; minimum; maximum) will be given for distorted data, and the number and percentage will be given for the representation of categorical variables.

In the comparison of numerical variables in the study groups, the appropriate method from the independent two-sample t-test and the Mann Whitney U test will be used by examining the necessary assumptions, and the Chi-square test for the comparison of categorical variables. Comparison of knowledge score before and after will be done with paired two-sample t-test or Wilcoxon tests, as appropriate.

IBM SPSS Statistics 21.0 (IBM Corp. Released 2012. IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp.) program will be used for statistical analysis and calculations. The statistical significance level will be accepted as p <0.05 for the hypotheses to be established bilaterally.

Data Collection Tools:

Data will be collected with the data collection form. The data colection form consist of five parts. 1. Introductory Information Form; 2. Sexual and Reproductive Health Knowledge Test; 3. Marriage Adjustment Scale; 4. The New Sexual Satisfaction Scale: The New Sexual Satisfaction Scale; 5. Sexual Self-Efficacy Scale:

ELIGIBILITY:
Inclusion Criteria:

* Can read and write
* No vision or hearing problems,
* Can use computer and internet,
* Expressing himself on the phone call,
* Those who have not received professional help due to any psychiatric or sexual dysfunction,
* Couples who have decided to get married

Exclusion Criteria:

* Couples with previous marital experience and who do not agree to work will not be included.
* Those diagnosed with psychiatric illness or sexual dysfunction after marriage will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
introductory information form | Baseline (pre-education)
  sociodemographic characteristics, marital characteristics
sexual and reproductive health knowledge level | Baseline (pre-education)
  It is a test consisting of 25 questions prepared by the researcher and scored between 0 and 100 pounds.

SECONDARY OUTCOMES:
sexual and reproductive health knowledge level | 1 month after marriage
  Test scored between 0-100 on sexual and reproductive health
sexual and reproductive health knowledge level | 4 months after marriage
  Test scored between 0-100 on sexual and reproductive health
Marital adjustment scale | 4 months after marriage
  Marital Adjustment Test; It measures the marital adjustment of married individuals.
  The scale consists of 15 items with different number of options. Each item gets a score between 0 and 6, which differs according to the number of options. According to this; 1st item 0-6 points, 2nd - 9. items 0--5 points, items 10 and 14 0--2 points, items 11 and 13 0--3 points, item 12 points if the option of sitting at home for one of the spouses and doing something outside for the other spouse is 0 points, each spouse The total score from the scale ranges from 0 to 60, with a score of 1 if the option to do something outside was selected, 2 points if the option to stay at home was selected for each spouse, and 0--2 points for the 15th item. Those who score above 43 are considered compatible in terms of marital relations, and those who score below are considered as incompatible.
New sexual satisfaction scale | 4 months after marriage
  New sexual satisfaction scale; It measures sexual satisfaction in women and men.
  The scale developed to measure sexual satisfaction in clinical and field studies is a 5-point Likert-type (1-5) measurement tool. The lowest score that can be obtained from the scale is 20, and the highest score is 100. The scale consists of the self-centered sub-dimension and the co-partner / sexual activity-centered sub-dimension. These two sub-dimensions represent the New Scale of Sexual Satisfaction. Self-centered subdimension 1-10. items, co-partner / sexual activity-centered sub-dimension 11-20. are substances. The new sexual satisfaction scale is items 1-20. The scoring of the scale is calculated by adding the items. Higher scores on the scale indicate good sexual satisfaction.
Sexual Self-Efficacy Scale | 4 months after marriage
  Sexual Self-Efficacy Scale; It measures the sexual self-efficacy of individuals.
  The scale is an 8-point Likert (0 Strongly Disagree - 8 Strongly Agree) type measurement tool consisting of 5 items with one factor. The scale gives total score. Items 3 and 4 of the scale are reverse coded. High scores indicate a high level of sexual self-efficacy. Possible score range that can be obtained from the scale is 0 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru İnan Kırmızıgül, Midwife, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Çankaya Vedat Dolakay Evlendirme Dairesi, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moodi M, Miri MR, Reza Sharifirad G. The effect of instruction on knowledge and attitude of couples attending pre-marriage counseling classes. J Educ Health Promot. 2013 Sep 30;2:52. doi: 10.4103/2277-9531.119038. eCollection 2013. PMID 24251288
- [Background] Vural BK, Temel AB. Effectiveness of premarital sexual counselling program on sexual satisfaction of recently married couples. Sex Health. 2009 Sep;6(3):222-32. doi: 10.1071/SH08065. PMID 19653960
- [Background] Puri S, Dhiman A, Bansal S. Premarital health counseling: A must. Indian J Public Health. 2016 Oct-Dec;60(4):287-289. doi: 10.4103/0019-557X.195860. PMID 27976650